CLINICAL TRIAL: NCT02573974
Title: Study of Alterations in Skeletal Muscle Energy Metabolism in Undernourished Patients With Gastrointestinal Cancer
Brief Title: Skeletal Muscle Energy Metabolism in Undernourished Patients With Gastrointestinal Cancer
Acronym: METERMUCADIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Inserm U1069 - Team Nutrition, Growth and Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PHAO14-TL/METERMUCADIG; 2015-A00683-46 (Registry Identifier: IdRCB); 2015-R25 (Other: CPP); 150963B-12 (Other: ANSM)
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Undernutrition; Gastrointestinal Cancer
Keywords: undernutrition; gastrointestinal cancer; skeletal muscle; energy metabolism
MeSH Terms: conditions — Malnutrition; Gastrointestinal Neoplasms | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case group (Other): the intervention, specific to the study, is to take samples on patients with advanced gastrointestinal cancer
  Interventions: Other: Samples
- Control group (Other): the intervention, specific to the study, is to take samples on non-undernourished patients supported for adjuvant chemotherapy as part of colorectal cancer
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Blood samples, muscle biopsy and sample of hair

SUMMARY:
Undernutrition associated with cancer, or cancer cachexia results from a deterioration of the energy balance that leads to a gradual mobilization of energy reserves in the body and to increasing deterioration of the nutritional status of patients. This will thus significantly reduce quality of life and survival of patients with a lower tolerance to cancer treatments. Despite undeniable progress in knowledge, many pathophysiological mechanisms remain few or not explored, which could explain that there is still no satisfactory therapeutic solution to halt the gradual deterioration of the nutritional status of patients. In this sense, apart from preclinical data obtained in animal models, there is currently no clinical study on the functioning of skeletal muscle energy metabolism in undernourished patients suffering of cancer.

ELIGIBILITY:
Case group selection criteria:

Inclusion Criteria:

* 18 years ≤ Age ≤ 80 years
* Colorectal pancreatic cancer
* Undernutrition related to cancer (weight loss > 5% weight in one month or 10% in 6 months)
* Indication to systemic chemotherapy
* Indication to the development of an implantable port
* Life expectancy ≥ 3 months
* WHO General Status ≤ 2
* Patients affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* Pregnant or breastfeeding women
* Unbalanced Diabetes
* Systemic corticosteroid treatment
* Any severe uncontrolled medical condition
* Alopecia

Control group selection criteria:

Inclusion Criteria:

* 18 years ≤ Age ≤ 80 years
* Colorectal pancreatic cancer
* Indication adjuvant chemotherapy
* Indication to the development of an implantable port
* Life expectancy ≥ 3 months
* WHO General Status ≤ 2
* Patients affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* Pregnant or breastfeeding women
* Undernutrition related cancer (weight loss > 5% weight in one month or 10% in 6 months)
* Unbalanced Diabetes
* Systemic corticosteroid treatment
* Any severe uncontrolled medical condition
* Alopecia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Measurement of muscle mitochondrial bioenergetics | An average of one week
  Measurement of muscle mitochondrial bioenergetics by high resolution oxygraphy

SECONDARY OUTCOMES:
Quantification of muscle lipid droplets | An average of one week
  Quantification of muscle lipid droplets by electron microscopy
Analysis of the expression of target genes and proteins | An average of one week
  Analysis of the expression of target genes and proteins involved in 1/ mitochondrial metabolism 2/ lipid metabolism 3/ the regulation of energy metabolism and 4/ muscle proteolysis by RTqPCR with SYBR Green and by Western Blot
Determination of body composition (fat mass / lean mass) | Within 4 weeks before inclusion
  Determination of body composition ( fat mass / lean mass ) by an imaging method scannographic
Determining the isotopic composition of nitrogen hair | An average of one week
  Determining the isotopic composition of nitrogen hair spectrometry .

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LECOMTE, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Service d'Hépato-gastroentérologie et de Cancérologie Digestive, CHRU de TOURS, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dolly A, Lecomte T, Tabchouri N, Caulet M, Michot N, Anon B, Chautard R, Desvignes Y, Ouaissi M, Fromont-Hankard G, Dumas JF, Servais S. Pectoralis major muscle atrophy is associated with mitochondrial energy wasting in cachectic patients with gastrointestinal cancer. J Cachexia Sarcopenia Muscle. 2022 Jun;13(3):1837-1849. doi: 10.1002/jcsm.12984. Epub 2022 Mar 22. PMID 35316572